CLINICAL TRIAL: NCT06926777
Title: Comparative Analysis of Median Nerve Parameters for Carpal Tunnel Syndrome (CTS) Diagnosis: Ultrasound Versus Nerve Conduction Studies (NCS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Combined Military Hospital Kohat Pakistan (Other Government)
Responsible Party: Principal Investigator, Syed Tameem Ul Hassan, Doctor, Combined Military Hospital Kohat Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: E-2005/A/114
Record Dates: First submitted 2025-03-15; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Carpal Tunnel Syndrome (CTS); Nerve Conduction; Ultrasound
Keywords: Carpal Tunnel Syndrome; Numbness; Tingling; Ultrasound; Nerve Conduction Study; Hand Weakness
MeSH Terms: conditions — Carpal Tunnel Syndrome; Hypesthesia; Paresthesia | interventions — Nerve Conduction Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound Diagnostic Arm (Other): Participants in this arm will undergo ultrasound imaging of the median nerve at the wrist. Measurements such as CSA and flattening ratio will be recorded. The goal is to evaluate ultrasound's effectiveness in diagnosing CTS compared to NCS.
  Interventions: Diagnostic Test: Nerve Conduction Study
- Nerve Conduction Study (NCS) Group (Diagnostic Arm) (Other): Participants in this arm will undergo an NCS to assess median nerve function. Parameters such as nerve conduction velocity, latency, and amplitude will be recorded. NCS findings will serve as the gold standard for comparison with ultrasound results.
  Interventions: Diagnostic Test: Nerve Conduction Study

INTERVENTIONS:
Diagnostic Test: Nerve Conduction Study — This study involves two diagnostic interventions for evaluating CTS:
  Ultrasound Examination (Diagnostic Intervention)
  1. A high-frequency ultrasound probe will be used to assess the median nerve at the wrist.
  2. Parameters measured include cross-sectional area, flattening ratio, and echogenicity.
  The goal is to determine if ultrasound can accurately diagnose CTS compared to NCS.
  NCS (Diagnostic Intervention)
  1. Surface electrodes will be placed on the skin to stimulate and record median nerve conduction.
  2. Parameters such as latency, conduction velocity, and amplitude will be recorded.
  3. NCS serves as the gold standard for diagnosing CTS and will be used for comparison with ultrasound results.
  Each participant will undergo both ultrasound and NCS, allowing researchers to compare their effectiveness in diagnosing CTS.

SUMMARY:
Comparative Analysis of Median Nerve Parameters for Carpal Tunnel Syndrome (CTS) Diagnosis: Ultrasound vs. Nerve Conduction Study (NCS) This clinical study aims to determine whether ultrasound can be as practical as NCS in diagnosing CTS. It will also evaluate the accuracy of different median nerve measurements in both tests.

The main questions it aims to answer are:

Can ultrasound accurately detect CTS compared to NCS? Which median nerve measurements (such as size, speed, or function) are most useful for diagnosis? Researchers will compare ultrasound and NCS results in patients with CTS symptoms to determine which test is more reliable and patient-friendly.

Participants will:

1. Undergo both an ultrasound and a NCS for comparison.
2. Visit the clinic for testing and evaluation as part of the study.
3. Provide information about their symptoms and medical history related to CTS. This study aims to improve diagnosis accuracy and explore whether ultrasound could be a more comfortable and quicker alternative to NCS for detecting CTS.

DETAILED DESCRIPTION:
This study aims to compare ultrasound and NCS for diagnosing CTS by analyzing key median nerve parameters in both tests. CTS is a common condition caused by compression of the median nerve at the wrist, leading to symptoms such as numbness, tingling, and weakness in the hand. Accurate diagnosis is essential to ensure appropriate treatment.

Currently, NCS is considered the standard test for CTS diagnosis, measuring nerve function by assessing conduction velocity and latency. However, ultrasound has emerged as a potential alternative by providing structural imaging of the median nerve, including parameters like cross-sectional area (CSA), echogenicity, and flattening ratio.

The primary objective of this study is to determine whether ultrasound can be a reliable, non-invasive, and patient-friendly alternative to NCS for CTS diagnosis. By comparing nerve measurements obtained from both methods, researchers aim to evaluate their diagnostic accuracy, sensitivity, and specificity.

Participants with suspected CTS will undergo both ultrasound and NCS for comparison. Data will be analyzed to determine which test provides the most precise and clinically useful information. The findings of this study may help refine diagnostic protocols, potentially reducing the need for NCS in certain cases and offering a faster, more comfortable option for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older.
2. Patients with clinical symptoms of CTS, including numbness, tingling, pain, or weakness in the hand.
3. Positive findings on clinical examination, such as Tinel's sign, Phalen's test, or Durkan's test.
4. Willingness to undergo both ultrasound and NCS for diagnostic evaluation.

Exclusion Criteria:

1. Previous surgery for CTS in the affected hand.
2. History of peripheral neuropathy such as diabetic neuropathy
3. Other neuromuscular disorders affecting the upper limb such as cervical radiculopathy.
4. Pregnant women.
5. Severe comorbid conditions that may interfere with study participation.
6. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Ultrasound Compared to Nerve Conduction Study for Carpal Tunnel Syndrome | Baseline
  Measuring the sensitivity, specificity, and overall accuracy of ultrasound in diagnosing CTS compared to NCS Parameters, including Median Nerve Latency, Amplitude, and Nerve Conduction Velocity

CONTACTS AND LOCATIONS:
Overall Officials: Syed Tameem Ul Hassan, MBBS, FCPS, Principal Investigator — Combined Military Hospital Kohat
Locations (1):
- Combined Military Hospital, Kohat, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Following IPD will be shared
  1. De-identified demographic data that is age, gender, relevant medical history.
  2. Ultrasound measurements of the median nerve such as CSA and flattening ratio.
  3. NCS results such as latency, conduction velocity and amplitude.
  4. Clinical assessment findings such as Tinel's sign, Phalen's test results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the completion of study, data will be provided on demand and will be available for 6 months post completion.
Access Criteria: Researchers will be given access. Data will be shared via email.